CLINICAL TRIAL: NCT03964467
Title: Investigation of Central Priming Prior to Training of the Upper Extremity in Chronic Stroke
Brief Title: Priming With tDCS: Expanding the Window of Recovery in Chronic Stroke
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of the Sciences in Philadelphia (Other)
Collaborators: Chapman University (Other); Moss Rehabilitation Research Institute (Other); Thomas Jefferson University (Other)
Responsible Party: Principal Investigator, Gregory Thielman, Professor of Therapy and Neuroscience, University of the Sciences in Philadelphia
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 06-0008
Record Dates: First submitted 2019-05-22; First posted 2019-05-28 (Actual); Last update posted 2023-02-06 (Actual); Status verified 2023-02

CONDITIONS: Upper Extremity Paresis
Keywords: stroke; upper extremity; intervention; transcranial direct current stimulation; actigraph; fMRI
MeSH Terms: conditions — Paresis; Stroke | interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Intervention Model Description: randomized controlled trial
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: PI is only doing the testing, while the trainers are training all the participants
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Experimental (Experimental): Transcranial Direct Current Stimulation.1) Scalp measurements of the scalp will be taken using the 10-20 EEG measurement system to determine anode and cathode placement. 2) One 1x1 Bicarbon electrode with wires attached will be placed in the center of each 5 cm x 7 cm sponge electrode dampened with 8 ml of saline. 3) One sponge electrode will be placed over the ipsilesional PMd (F3) and the other sponge electrode over the contralesional supraorbital region(Fp2). 4) Each sponge electrode will be secured under the plastic EZ strap 5) The current from the Actividose II will be turned up to 2 MA. The current will ramp up/down in 15 seconds. We will observe for adverse effects and hit the pause button, then turn the machine off, if a participant does not tolerate the stimulation. Individuals in this arm will have the stimulation stay in current until the full dose is delivered. Each participant will then engage in the UE TRT as outlined below.
  Interventions: Device: transcranial direct current stimulation
- Control (Sham Comparator): Individuals in this arm will have the stimulation cycled off after 2-3 minutes. All will be part of the Circuit-Based, UE Task Related Training. Each participant will engage in the training program for 1.5 hours; rotating through 5 stations at about 15 minute intervals, participating in standing as tolerated, but stations can be adapted to sitting. The goal is for each participant perform > 225 movements with the affected arm per session, at the highest functional level. Rest breaks given as needed. Examples of stations are: Reach-to-grasp tasks to objects of various weight, texture and dimension at different distances and table heights. Practice opening simulated locks and containers. Shoulder wheel involving grasping plastic plates with varied grip patterns and sliding them up and over the wheel from the unaffected to the affected side encouraging shoulder abduction, external rotation and supination. Bimanual/unimanual ball toss: catching, releasing.
  Interventions: Device: transcranial direct current stimulation

INTERVENTIONS:
Device: transcranial direct current stimulation — see arm/group descriptions
  Other Names: Upper extremity Circuit training

SUMMARY:
Stroke often leads to long-term disability including upper extremity (UE) dysfunction even with the provision of timely rehabilitation services. Brain injury stemming from stroke, affecting the corticospinal system results in weakness, alterations in muscle tone and incoordination during the performance of functional tasks. Recovery of functional task performance after injury to the corticospinal system involves a residual neural network that engages the premotor cortex, frontal cortex and supplementary motor cortex. In particular, the dorsal premotor cortex (PMd) is anatomically and physiologically poised to reorganize and support motor recovery after corticospinal damage. The goal of this study is to determine the feasibility and efficacy of stimulating the ipsilesional PMd in adults with chronic stroke using noninvasive anodal transcranial direct current stimulation (tDCS) during the training sessions of a 4-week circuit-based, UE, task-related training (TRT) program. Pilot data from six adults, using anodal tDCS over the injured PMd just before each session of TRT, led to significant improvements in UE function in 5 of the 6 adults after only 4 weeks of training. We will assess the motor function of both arms using clinical assessments immediately before and after the 4-week TRT program. In addition to effects of tDCS-primed UE-TRT on clinical outcomes, we will use functional magnetic resonance imaging (fMRI) to determine the changes in neural network reorganization. We hypothesize that the training program will reveal significant improvement in motor function based on clinical assessment as well as significant global network changes based on resting state functional MRI and hybrid diffusion MR imaging. The long-term goal of this research is to develop an effective intervention strategy to improve UE function in individuals with moderate impairment from chronic stroke.

DETAILED DESCRIPTION:
AIM 1: To determine if UE motor performance significantly improves in individuals with moderate impairment from chronic stroke, following anodal tDCS applied to the ipsilesional PMd during circuit-based, UE, TRT conducted three times/week for 4-weeks. Hypothesis: Following a 4-week, tDCS-paired UE TRT program, there will be significant changes in unimanual and bimanual performance in individuals with moderate impairment from chronic stroke, as detected by clinical assessments. Our primary measure will be UE accelerometry gathered with wrist-based ActiGraphs; a secondary measure will be the Wolf Motor Function Test (WMFT).

AIM 2: To determine if there are significant structural and functional brain changes in individuals with moderate impairment from chronic stroke, following anodal tDCS applied to the ipsilesional PMd paired with circuit-based, UE, TRT conducted 3 times/week for 4-weeks. Hypothesis: Following a 4-week, tDCS-paired UE TRT program, there will be significant structural/functional brain changes as detected by magnetic resonance imaging (MRI) and functional MRI (fMRI). Based on prior work,4,10 we expect that there will be an increase in resting state functional connectivity as shown using BOLD fMRI between the cerebellum and cortical areas.

Task related training (TRT) is a treatment approach that aims to increase use of the paretic arm, avoid learned disuse and minimize compensation (Thielman et al, 2004). It involves variable practice of goal-directed, functional movements in a natural environment (Ada et al, 1994) focusing on solving movement problems (Gentile, 2000). Task related training has been found to significantly improve paretic arm function post-stroke, in individuals with baseline UE FM < 35 (Kim et al., 2013; Thielman et al., 2004; Thielman, 2015; Wu et al, 2000).

The effects of TRT could be augmented with noninvasive brain stimulation pairing. Motor priming before or during task practice has been found to foster motor learning and UE function in healthy individuals and persons post-stroke by increasing neuroplasticity (Fusco et al., 2014; Stoykov and Madhavan, 2015; Stoykov and Stinear, 2010). Anodal transcranial direct current stimulation (tDCS) is one form of stimulation (Fusco et al., 2014). Anodal tDCS increases neuronal excitability by depolarizing the membrane potential while cathodal tDCS decreases excitability and hyperpolarizes the membrane potential (Nitsche and Paulus, 2001). After effects from anodal tDCS stimulation, involving activation of NDMA receptors associated with long-term potentiation, have been shown to last up to 120 minutes (min) (Madhavan and Shah, 2012). Anodal tDCS administered during intervention has a greater impact on UE function than therapy or tDCS alone (Bolognini et al., 2011; Butler et al., 2013; Cho et al., 2015; Lee and Lee, 2015; Yao et al., 2015). While the receipt of tDCS during therapeutic interventions is promising, it can limit the therapy to seated or more sedentary programs. Given the support in the literature, we believe it may be more effective to foster neuroplasticity and UE functional recovery in chronic stroke survivors if tDCS is done repetitively, during participation in a dynamic UE standing program. Our circuit-based, UE TRT standing program requires more aerobic effort from participants than seated programming and greater aerobic effort has been shown to foster neuroplasticity in persons post-stroke (Mang et al., 2013; Quaney et al., 2009).

Expanding Plasticity Beyond the Motor Cortex. The dorsal premotor cortex (PMd) may be a more suitable neural substrate for promoting recovery in moderately impaired individuals. While the results of anodal priming over the ipsilesional motor cortex are promising, the effects have primarily been limited to persons with mild impairments. For persons with moderate impairment, a substantial portion of the motor cortex and/or corticospinal system is damaged leaving less neural substrate within M1 than can be targeted using anodal tDCS. In such individuals, alternative cortical sites may have greater potential to reorganize and implement motor recovery. Previously, we (Kantak et. al., 2012) and others (Plow et al., 2016) proposed that the PMd may be uniquely poised to reorganize and implement recovery after motor cortex injury. The PMd contributes to over 30% of descending corticospinal fibers (Barbas and Pandya, 1987; Dum and Strick, 2002). Further, the PMd has been shown to reorganize after stroke, contributing to motor performance (Fridman et al., 2004; Kantak et al., 2012; Mohapatra et al., 2016). We believe that the benefit of priming the PMd before engaging in circuit-based, UE TRT warrants further investigation.

Brain Imaging. Using hybrid diffusion magnetic resonance imaging (MRI) and functional MRI (fMRI) to quantify structural and functional changes in the brain is critical to understand behavioral change post-injury and with training. Functional organization of intact cortical tissue post-stroke is dependent on the post-injury behavioral experience (O'Shea et al, 2007). Neuroimaging has been used to show an increase in neural activity in persons who engage in TRT post-stroke (Nelles et al,2001). By using fMRI to assess brain function, the volume of activation in regional brain areas can be determined, which could be used to predict treatment outcome (Cramer, 2008).

ELIGIBILITY:
Inclusion Criteria:

1. > 18-75 years of age;
2. diagnosis of ≥ 1 stroke > 6 months before participation;
3. in good health;
4. classified with moderate impairment based on the UE Fugl Meyer Assessment (FMA; score of 19-47
5. safe for the MRI environment;
6. able to elevate and hold the paretic arm for 2 seconds at 90 degs shoulder elevation, 160-180O elbow extension and neutral forearm supination;
7. ≥ 20 degrees gravity minimized wrist extension while holding a cylindrical object on a tabletop.

Exclusion Criteria:

1. bone or joint limitations that restrict paretic arm motion;
2. history of skull fractures or burr hole(s);
3. resting heart rate and resting blood pressure outside the range of 40-100 beats/min and 90/60 to 170/90 mm Hg respectively;
4. chest pain or shortness of breath at rest;
5. history epilepsy or seizures;
6. Botox injections to the paretic arm within 4 months of participation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2019-01-14 (Actual); Primary Completion 2023-04-14 (Estimated); Study Completion 2023-04-14 (Estimated)

PRIMARY OUTCOMES:
UE Accelerometry | 3 day period prior to training
  actigraph markers placed on each arm
UE Accelerometry | 3 day period post training to assess change- more activity inbdicates greater overall use
  actigraph markers placed on each arm
Functional MRI | within 3 days prior to training
  fMRI consisting of structural data collected, DTI, resting state data functional task data
Functional MRI | within 3 days post training to measure change- increased activity in designated areas explains pattern of neuroplasticity
  fMRI consisting of structural data collected, DTI, resting state data and functional task data

SECONDARY OUTCOMES:
Body Structure Function and Impairment Data | 1-3 days prior to training start
  Impairment measures- FMA
Body Structure Function and Impairment Data | 1-3 days post training
  Impairment measures- FMA (19-47. with higher scores indicating positive change)
Body Structure Function and Impairment Data | 1-3 days prior to training start
  Impairment measures- grip strength (0-60 Kg, with higher scores indicating increased strength
Body Structure Function and Impairment Data | 1-3 days post training
  Impairment measures- grip strength
Body Structure Function and Impairment Data | 1-3 days prior to training start
  Impairment measures- AROM
Body Structure Function and Impairment Data | 1-3 days post training
  Impairment measures- AROM (elbow extension- minus 30 to 0, with 0 being full positive for full extension; shoulder flexion- 90 - 180, with greater excursion indicating greater positive progress
Body Structure Function and Impairment Data | 1-3 days prior to training start
  Activity measures-Wolf Motor Function Test- time to complete task
Body Structure Function and Impairment Data | 1-3 days post training
  Activity measures-Wolf Motor Function Test- time to complete task indicated- with less time indicting improvement
Body Structure Function and Impairment Data | 1-3 days prior to training start
  Patient Reported measure- Stroke Impact Scale-
Body Structure Function and Impairment Data | 1-3 days post training
  Patient Reported measure- Stroke Impact Scale- pt.reports changes on named activities participation in real world on a 1-5 point Likert scale across the 8 domains, with higher scores indicating less difficulty on the tasks

CONTACTS AND LOCATIONS:
Overall Officials: Gregory Thielman, EdD, Principal Investigator — Professor
Locations (1):
- University of the Sciences, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Yes
all fMRI data will be made available to the ENIGMA Stroke group as a member of this consortium.
  The behavioral data is available publicly as able on this or any site I am directed to. Often I am contacted individually by the PI of systematic reviews for this type of data
Supporting Information: Study Protocol, SAP, ICF
Time Frame: as requested and up to 5 years